CLINICAL TRIAL: NCT01575327
Title: Using a Closed-loop System for Oxygen Delivery (FreeO2) to Optimize Exercise Tolerance During Walk in Patients With COPD, Oxygen Therapy and Hypercapnia
Brief Title: Closed-loop System for Oxygen Delivery and Exercise in Chronic Obstructive Pulmonary Disease
Acronym: FreeO2-rehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AGIR à Dom (Other)
Collaborators: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 11-AGIR-01
Record Dates: First submitted 2012-03-13; First posted 2012-04-11 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2017-01

CONDITIONS: COPD; Oxygen Therapy; Hypercapnia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypercapnia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fixed oxygen flow delivery (Active Comparator): Oxygen flow delivery is adjusted by respiratory therapists. Standard medical treatment.
  Interventions: Device: Manual settings with FreeO2 system in collection mode
- FreeO2 system (Experimental): FreeO2 is a new system that automatically adjusts the oxygen flow delivered to patients in a closed-loop based on the SpO2 signal. This system is intended to maintain SpO2 in a predefined target and to adapt oxygen flow to patient's needs.
  Interventions: Device: Automated settings on the oxygen delivery device

INTERVENTIONS:
Device: Automated settings on the oxygen delivery device — FreeO2 automatically adjusts the oxygen flow delivered to patients based on the SpO2 signal and collects the cardiorespiratory parameters
  Arms: FreeO2 system
Device: Manual settings with FreeO2 system in collection mode — FreeO2 system does not adjust oxygen flow but collects the cardiorespiratory parameters
  Arms: Fixed oxygen flow delivery

SUMMARY:
The purpose of this study is to investigate the benefit of Closed-loop System for Oxygen Delivery (FreeO2) as compared with fixed oxygen flow during endurance shuttle walking test in patients with Chronic obstructive pulmonary disease (COPD), oxygen therapy and hypercapnia.

The study was designed to test the following hypotheses:

As compared with fixed oxygen flow, the FreeO2 Oxygen Delivery system leads to higher exercise tolerance (distance during ESWT) and lower desaturation events without increase in hypercapnia in patients with COPD, oxygen therapy and hypercapnia.

As compared with fixed oxygen flow, the FreeO2 Oxygen Delivery system leads to lower dyspnea and leg fatigue scores at a given endurance time during the shuttle walking test in patients with COPD, oxygen therapy and hypercapnia.

As compared with fixed oxygen flow, the FreeO2 Oxygen Delivery system leads to lower cardiac and respiratory frequencies at a given endurance time during the shuttle walking test in patients with COPD, oxygen therapy and hypercapnia.

DETAILED DESCRIPTION:
Background:

In spite of oxygen therapy, desaturations frequently occur during exercise in COPD patients. Although current recommendations are to add 1 L/min to the baseline oxygen flow during exertion, a new closed-loop system (FreeO2) automatically and continuously adjusts the oxygen flow to the patient's needs based on the oxygen saturation by pulse oximetry (SpO2), end-tidal CO2 (EtCO2) and respiratory rate. A preliminary study showed significant improvement in exercise tolerance in COPD patients not needing oxygen therapy. Although oxygen flow could be two fold increased during exercise, a worsening hypercapnia is plausible in severe COPD.

Aim of this study is to evaluate this system during endurance shuttle walking test in COPD patients with oxygen therapy and hypercapnia.

Methods: The investigators proposed to conduct a controlled, randomized cross-over study comparing the efficacy of a Closed-loop System for Oxygen Delivery (FreeO2) as compared with fixed oxygen flow during an endurance shuttle walking test in patients with COPD, oxygen therapy and hypercapnia.

ELIGIBILITY:
Inclusion Criteria:

* 40 Years and older
* Patient with COPD severe to very severe requiring long-term Oxygen Therapy
* Hypercapnia (PaCO2 > 45mmHg)
* Former or current smoker greater than or equal to 10 pack-years

Exclusion Criteria:

* Pregnant or breast-feed woman
* Patients under guardianship
* Imprisoned patients

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in Endurance time | Day 0 (inclusion) + 14 and D0 +21
  Duration during the endurance shuttle walking test

SECONDARY OUTCOMES:
Change in Dyspnea during ESWT | Day 0 (inclusion) + 14 and D0 +21
  Visual analogic scores of dyspnea during the endurance shuttle walking test
Change in Muscle fatigue during ESWT | Day 0 (inclusion) + 14 and D0 +21
  Visual analogic scores of leg discomfort during the endurance shuttle walking test
Change in Respiratory frequency during ESWT | Day 0 (inclusion) + 14 and D0 +21
  Respiratory frequency measurement by the FreeO2 system during the endurance shuttle walking test
Change in PaCO2 during ESWT | Day 0 (inclusion) + 14 and D0 +21
  EtCO2 measurement by the FreeO2 system during the endurance shuttle walking test
Hypercapnia level at baseline | Day 0 (inclusion) - baseline evaluation
  Blood gases at rest
Change in Cardiac frequency during ESWT | Day 0 (inclusion) + 14 and D0 +21
  Cardiac frequency measurement by the FreeO2 system during the endurance shuttle walking test
Change in SpO2 during ESWT | Day 0 (inclusion) + 14 and D0 +21
  Pulse oxygen saturation during the endurance shuttle walking test

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Pepin, MD, PhD, Principal Investigator — Laboratoire EFCR, CHU de Grenoble, 38043, Grenoble, France
Locations (3):
- France (3):
  - Hopital Universitaire, Grenoble
  - Centre ATRIR, Nyons
  - Centre Henri BAZIRE, Saint-Julien-de-Raz

REFERENCES:
- [Derived] Vivodtzev I, L'Her E, Vottero G, Yankoff C, Tamisier R, Maltais F, Lellouche F, Pepin JL. Automated O2 titration improves exercise capacity in patients with hypercapnic chronic obstructive pulmonary disease: a randomised controlled cross-over trial. Thorax. 2019 Mar;74(3):298-301. doi: 10.1136/thoraxjnl-2018-211967. Epub 2018 Aug 30. PMID 30166425